CLINICAL TRIAL: NCT03309527
Title: A Double-blind Randomized Controlled Study on Influence of E-aid Cognitive Behavioral Therapy for Insomnia to Reduce Incidence of Depression as Well as Suicidal Ideation in Patients With Insomnia
Brief Title: E-aid Sleep-focused TrEatment for Prevention of Major Depression (STEP-MD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NFEC-2017-132
Record Dates: First submitted 2017-09-25; First posted 2017-10-13 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Insomnia; Depression; Self Harm
Keywords: insomia; Depression; Self Harm; Suicide; guided self-help; psychological treatment; eCBTI; internet; Psychotherapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression; Self-Injurious Behavior; Suicide

STUDY DESIGN:
Intervention Model Description: A two-arm parallel design involves two groups of participants with insomnia. One group receives internet delivered sleep hygiene education, and the other group receives internet delivered cognitive behavior therapy.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-aid Cognitive Behavior Therapy (Experimental): Participants receive e-aid cognitive behavior therapy. Every week, this group will receive researcher guided individual customized sleep restriction and stimulus control therapy.
  Interventions: Behavioral: e-aid Cognitive Behavior Therapy
- e-aid Sleep Hygiene Education (Active Comparator): Participants receive e-aid sleep hygiene education which consists of general sleep health education and the guidance on questionnaires. Every week, this group will receive researcher guided sleep hygiene.
  Interventions: Behavioral: e-aid Sleep Hygiene Education

INTERVENTIONS:
Behavioral: e-aid Cognitive Behavior Therapy — e-aid Cognitive Behavior Therapy
  Arms: e-aid Cognitive Behavior Therapy
Behavioral: e-aid Sleep Hygiene Education — e-aid Sleep Hygiene Education
  Arms: e-aid Sleep Hygiene Education

SUMMARY:
In the past, there were studies on relationship between insomnia and depression, and those studies found that depression can be the result of untreated insomnia. Mostly insomnia precedes depression, and is a marker for recurrence of depression. Research suggests that insomnia may cause depression by changing the emotional response.

In this study, investigators will establish the national online cognitive behavioral therapy for insomnia (e-aid Cognitive Behavioral Therapy for Insomnia, eCBTI ) tools, and online health education on sleep (e-aid Sleep Hygiene Education, eSHE ) tools for controls. Investigators will be testing whether eCBTI can reduce the incidence of depression in patients with sleep disorders, increasing remission rate of depression, and a corresponding reduction in suicidal ideas, compared with eSHE control groups.

DETAILED DESCRIPTION:
1000 patients suffering from insomnia will be recruited in this study.Participants with insomnia will be taken from: A. the WeChat platform, B. the customer group of intelligent hardware/software, and C.outpatient department. 1000 participants with insomnia will be randomly divided into eCBTI group and eSHE group equally that each group will have 500 participants.

Participants will be requested to accept online structured questionnaire, including social and demographic data and insomnia disorders diagnosis process (adapted from "A guide to diagnosis and treatment of insomnia in China"). If the interviewee meets the criteria of entry, then participants are requested to fill online informed consent and then enrolled into the baseline assessment.

Baseline assessment includes two parts:

1, Self-reported questionnaire: Insomnia Severity Index, ISI, Dysfunctional Beliefs and Attitudes about Sleep, DBAS, Sleep Hygiene and Practices Scale, SHPS, Pre - Sleep Arousal Scale, PSAS, Epworth Sleepiness Scale, ESS, Hospital Anxiety and Depression Scale, HADS, Short - Form 12 - Item Health Survey, SF - 12; 2. Researcher Interview: Clinical Interview of depression in the Mini International Neuropsychiatric Interview (MINI).

Therapeutic intervention: Both groups will be treated for 4 weeks, and multiple follow-up visits within 12 months.

The research specifically tailored the third-party application of the smartphone to complete the online insomnia therapy program. The eCBTI group and the eSHE group included four weeks of core courses: daily listening to five minutes of sleep hygiene education, and recording sleep diaries. Every week, eCBTI group will receive guided individual customized sleep restriction and stimulus control therapy whereas eSHE group will be given sleep health education and the guidance regarding questionnaires.

Previous studies have shown that the annual prevalence of depression in people with insomnia is about 2 to 3 percent. Based on investigators previous research results, new cases of depression were 7.4%, and patients with chronic insomnia eCBTI treatment can effectively reduce the depression incidence rate by 50%, such as the need to achieve 80% Confidence Interval at p-value of 0.05, 300 patients will be needed in each group. Considering the loss rate of about 30-40%, the study required 500 cases per group (eCBTI group and eSHE group) in the baseline.

Outcomes will be measure in continuous variable data with mean and standard deviation (SD), classifying data with numerical value or percentage. Compare parametric data and non-parametric data (2 groups) through independent t-test. The variance analysis of repeated measures will be used to compare the difference between the two groups in treatment and follow-up (e.g., ISI, etc.). The 2 classification variables of clinical results will be calculated by survival analysis, such as the new suicidal thoughts in two groups. Bilateral 5% significance level is statistically significant. All statistical programs are implemented in the 22.0 version of the social science statistical package (IBM SPSS 22.0) that runs in Windows.

ELIGIBILITY:
Inclusion Criteria:

* the diagnostic criteria for insomnia in accordance with DSM-5
* 18 years or older
* compliant and have a good understanding of research program
* able to fill the online informed consent form
* owns and have a good command on electronic gadgets (e.g., smart phones, tablets, computers, etc.)

Exclusion Criteria:

* clear and unhealed physical, mental and/or sleep disorders requiring acute care
* is taking psychotherapy for insomnia
* shift workers, regular night shift workers, frequent time zone fliers (such as crew members on international flights)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
occurrence of depression | changes of occurrence of depression from baseline to 2weeks, 5 weeks, 6 months and 12 months.
  Clinical Interview of depression in the Mini-International Neuropsychiatric Interview (MINI) by investigators by telephone or online.

SECONDARY OUTCOMES:
Treatment adherence rating scale | changes of scale score from baseline to 6 months and 12 months
  A self-reported questionnaire will be administered posttreatment to assess adherence to CBTI guidelines and the perceived helpfulness of treatment guidelines. Adherence to each therapeutic element will be rated on a 0 to 3 scale as follows: (0) Followed rarely or not at all; (1) Followed occasionally; (2) Followed most of the time; (3) Followed consistently. Ratings for all therapeutic elements will be broadly grouped into a Behavioral Component and a Cognitive Component. The Behavioral Component consists of stimulus control and sleep restriction guidelines and will include the following 4 items: adhering to a fixed prescribed bedtime, getting out of bed when unable to sleep, using the bed only for sleep, and restricting the amount of time spent in bed (Cronbach α = 0.50). The Cognitive Component consists of endorsement of 2 items: "Changing my expectations about sleep" and "Changing the way I think about not sleeping" (Cronbach α = 0.83)
Treatment satisfaction rating scale (TSRS) | changes of scale score from baseline to 6 months and 12 months
  Subjects' satisfaction to the treatment measured by Treatment satisfaction rating scale.The Consumer Report Treatment satisfaction scale will be adapted for insomnia in the study as: "How much do you feel the insomnia treatment program has helped you in the following areas?" The areas will include insomnia, energy level, work productivity, coping, life enjoyment, hopefulness, self-esteem, and mood. Each item will be rated on a 5 point Likert scale, with 1 = Made things a lot better; 2 = Made things somewhat better; 3 = Made no difference; 4 = Made things somewhat worse; 5 = Made things a lot worse. All items on this measure will be coded such that higher scores indicates greater symptom improvement. Overall treatment satisfaction was computed as the average score on all 7 items of the TSRS, which provided an index of clinically significant improvement (Cronbach α = 0.86).
Changes in Insomnia Severity Index(ISI) | changes of scale score from baseline to 2 weeks, 5 weeks, 6 months and 12 months.
  The ISI is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia in the last month. The dimensions evaluated are: severity of sleep onset, sleep maintenance, and early morning awakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime functioning, noticeability of sleep problems by others, and distress caused by the sleep difficulties. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28. The internal consistency of the ISI was found to be excellent (Cronbach's = 0.74) and has been validated with both sleep diary and polysomnography. This outcome will be measured at 2 weeks, 5 weeks, 6 months and 12 months in both the eCBTI and eSHE groups.
Changes in Hospital Anxiety and Depression Scale (HADS) | changes of scale score from baseline to 2 weeks, 5 weeks, 6 months and 12 months.
  The HADS is a self-report questionnaire to determine the levels of anxiety and depression that a participant is experiencing. The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression.Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. The HADS uses a scale and therefore the data returned from the HADS is ordinal. A cut-off point of 8/21 for anxiety or depression will be used. For anxiety (HADS-A) this gave a specificity of 0.78 and a sensitivity of 0.9. For depression (HADS-D) this gave a specificity of 0.79 and a sensitivity of 0.83.This outcome will be measured at 2 weeks, 5 weeks, 6 months and 12 months in both the eCBTI and eSHE groups.
Changes in Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS) | changes of scale score from baseline to 2 weeks, 5 weeks, 6 months and 12 months.
  The DBAS is a 30-item self-report questionnaire designed to evaluates sleep-related beliefs, querying respondents' expectations and attitudes regarding the causes, consequences, and potential treatments of sleep issues. The 30-item version showed adequate psychometric properties as evidenced by good internal consistency (Cronbach Alpha = 0.80), moderate item-total correlations (mean rs = 0.37), and adequate convergent and discriminant validity.Likert-type scale requiring participants to choose from 0 (strongly disagree) to 10 (strongly agree) will be used. Thus, the results are quantified in terms of strength of endorsed beliefs. A higher score indicates more dysfunctional beliefs and attitudes about sleep. The total score is based on the average score of all items.
Changes in Short - Form 12 - Item Health Survey（SF-12） | changes of scale score from baseline to 2 weeks, 5 weeks, 6 months and 12 months.
  The SF-12 is a 12-item self-report questionnaire used to assess generic health outcomes from the patient's perspective.The SF-12 addresses the 8 domains viz. Physical functioning (PF), Role - physical (RP),Bodily pain (BP),General health perceptions (GH),Vitality (V),Social functioning (SF),Role - emotional (RE) and Mental health (MH) . The 2 scores that will be obtained from this assessment are composite scores representing physical health and mental health composite summaries, PCS and MCS respectively. An algorithm will be used to generate the physical and mental health composite scores for comparison to normative data. In normative data, the mean score is set to 50, thus scores > 50 indicate better physical or mental health than the mean and scores < 50 indicate worse health.
Changes in Sleep Hygiene and Practices Scale(SHPS) | changes of scale score from baseline to 2 weeks, 5 weeks, 6 months and 12 months.
  Subjects' general sleep hygiene and practices are measured with Sleep Hygiene and Practices Scale.The SHPS is a 13-item self-report measure designed to assess the practice of sleep hygiene behaviors. Each item is rated on a five-point scale ranging from 0 (never) to 4 (always). Total scores range from 0 to 52, with a higher score representing poorer sleep hygiene. SHPS has shown adequate reliability and validity .
Changes in Pre-Sleep Arousal Scale(PSAS) | changes of scale score from baseline to 2 weeks, 5 weeks, 6 months and 12 months.
  Participant's problems during initiation of sleep is assessed with Pre-Sleep Arousal Scale.The Pre-Sleep Arousal Scale (PSAS) is a brief self-administered measure in which participants rate the intensity of experienced arousal. Internal consistency for somatic (8 items) and cognitive (8 items) subscales are satisfactory (α = 0.81 and α = 0.76) respectively.
Changes in Epworth Sleepiness Scale(ESS) | changes of scale score from baseline to 2 weeks, 5 weeks, 6 months and 12 months.
  Subjective measure of a patient's sleepiness is measured with Epworth Sleepiness Scale.The Epworth Sleepiness Scale is a self-report 8-item questionnaire producing scores from 0 to 24. Scores greater than 10 suggest significant daytime sleepiness. The Epworth Sleepiness Scale has good psychometric properties , correlates with objective measures of sleepiness , and has been shown to differentiate between individuals with and without sleep disorders and those who are and are not sleep deprived.
occurrence of suicidal ideation | changes of occurrence of suicidal ideation from baseline to 2 weeks, 5 weeks, 6 months and 12 months.
  Clinical Interview of suicidal ideation in the Mini-International Neuropsychiatric Interview (MINI) by investigators by telephone or online.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Zhang, MD & PhD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided